CLINICAL TRIAL: NCT05785377
Title: Efficacy of Neostigmine as an Adjuvant to Bupivacaine in Ultrasound-guided Transversus Abdominis Plane Block as a Postoperative Analgesia After Caesarean Delivery.
Brief Title: Neostigmine as an Adjuvant in Tranversus Abdominis Plane (TAP) Block in Cesarean Section Under Spinal Anesthesia
Acronym: TAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TAP-neostigmine
Record Dates: First submitted 2022-03-28; First posted 2023-03-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: according to the computer-generated random number codes that will be placed in sealed envelopes, the patients will be randomly allocated into two groups; Group-B and Group-BN according tho the local anesthetic injected in Ultrasound-guided bilateral Tranversus abdominis plane block
Who Masked: Participant, Investigator
Masking Description: The injectate used for TAPB will be prepared according to the group by an anesthesiologist who won't be involved in the data collection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine group (Group-B) (Placebo Comparator): After cession section, patients Will receive ultrasound (US)-guided bilateral TAP block with 20 mL bupivacaine 0.25% plus 1 mL of normal saline (Total volume of 21mL in each side
  Interventions: Drug: Bupivacaine
- Bupivacaine-Neostigmine group (Group-BN) (Active Comparator): After cession section, patients Will receive ultrasound (US)-guided bilateral TAP block with 20 mL bupivacaine 0.25% plus 1 mL of 500 mcg neostigmine (Total volume of 21mL in each side
  Interventions: Drug: Bupivacaine-Neostigmine

INTERVENTIONS:
Drug: Bupivacaine-Neostigmine — 20 mL bupivacaine 0.25% plus 1 mL Neostigmine (500 mcg)
  Arms: Bupivacaine-Neostigmine group (Group-BN)
Drug: Bupivacaine — 20 mL bupivacaine 0.25% plus 1 mL normal saline 0.9%
  Arms: Bupivacaine group (Group-B)

SUMMARY:
Cesarean birth is a common surgical procedure. After cesarean birth, postsurgical pain may delay recovery, interfere with maternal-newborn bonding, and reduce the breastfeeding if not adequately controlled. Postpartum analgesia has become a common concern.

Many adjuvant drugs used for peripheral nerve blocks as( N-methyl-d-aspartate (NMDA) receptor antagonists , Magnesium , Ephedrine , Dexamesathone , Fentanyl , Midazolam and Neostigmine) The potential of neostigmine as an adjuvant in peripheral nerve block is through its action to increase acetylcholine at muscarinic junctions of peripheral nerves. 500 mcg neostigmine was used as adjuvant to local anesthetic in an axillary brachial plexus block leads to decreased pain and less use of analgesics in the first 24 hours postoperatively with no incidence of adverse effects.

DETAILED DESCRIPTION:
This prospective double-blinded randomized controlled study will be done on parturients that are scheduled for elective cesarean delivery under spinal anesthesia to assess the efficacy of neostigmine as an adjuvant to isobaric bupivacaine inTranversus abdominis plane (TAPB) for postoperative analgesia in cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 40 years old
* American Society of Anesthesiologists (ASA) physical status II patients
* Singleton pregnancies with a gestational age of at least 37 weeks.
* Patients undergoing spinal anesthesia for cesarean delivery via a Pfannenstiel incision with exteriorization of the uterus.

Exclusion Criteria:

* Age < 19 or > 40 years.
* Height<150 cm, weight < 60 kg, body mass index (BMI) ≥40 kg/m2.
* Inability to comprehend or participate in the pain scoring system.
* Contraindications to spinal anesthesia (Coagulopathy, increased intracranial pressure, or local skin infection).
* Hypersensitivity to any drug used in the study.
* Any hypertensive disorders of pregnancy.
* Renal impairment or other contraindications to non-steroidal anti-infilamatory drugs (NSAIDS).
* Significant cardiovascular, renal or hepatic abnormalities.
* Patients with history of opioid intake, drug abusers or psychiatric patients

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — singleton pregnant women with a gestational age of at least 37 weeks
Enrollment: 58 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
The time of the first postoperative analgesic requirement | during the first 24 postoperative hours
  during the first 24 postoperative hours

SECONDARY OUTCOMES:
Total amount of the postoperative analgesic drugs (ketolac, paracetamol and fentanyl) consumed in the | during the first 24 postoperative hours
  mg
The visual analog scale (VAS) scores during rest | during the first 24 postoperative hours
  11-point VAS (where 0 for no pain and 10 for the worst possible pain) at 0, 2, 4,6,12 and 24 hours postoperatively
The visual analog scale (VAS) scores during movement | during the first 24 postoperative hours
  11-point VAS (where 0 for no pain and 10 for the worst possible pain) at 0, 2, 4,6,12 and 24 hours postoperatively
Mean arterial blood pressure (MBP) | basal (preoperative), intraoperative each 10 minutes and postoperatively every hour during first 6 hours
  mmHg
heart rate (HR) | basal (preoperative), intraoperative each 10 minutes and postoperatively every hour during first 6 hours
  beat per minute
Patient satisfaction about the quality of postoperative analgesia | during the first 24 postoperative hours
  poor = 1, fair = 2, good = 3, excellent = 4
The side effects (nausea, vomiting, abdominal colic and lower limb weakness) | during the first 24 postoperative hours
  incidence
the time from intrathecal injection till regression of spinal anesthesia to L2 dermatome | during the first 24 postoperative hours

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University-Emergency hospital-ICU, El Mansoura, Mansoura, Egypt